CLINICAL TRIAL: NCT01432028
Title: Polymorphisms in Genes Encoding the Estrogen Metabolism Enzymes and Effects of Hormone Therapy for Oral Low Dose or Not Oral on Variables Related Endothelial Function, Inflammation and Metabolic Profile in Patients in Recent Menopause Study Pharmacogenetic
Brief Title: Pharmacogenetic Study of Different Hormone Therapies in Recent Menopause Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denusa Wiltgen (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor-Investigator, Denusa Wiltgen, MD,PhD, Federal University of Rio Grande do Sul
Organization: Federal University of Rio Grande do Sul (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 05053
Record Dates: First submitted 2011-04-19; First posted 2011-09-12 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Postmenopause
MeSH Terms: interventions — Estradiol; Progesterone; drospirenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-oral hormone therapy (Active Comparator): 3 mg/day intranasal estradiol daily or 1,5 mg/day transdermal estradiol and 200 mg/day vaginal micronized progesterone for 14 days/month
  Interventions: Drug: Estradiol and Progesterone
- oral homone therapy (Active Comparator): estradiol 1mg and drospirenone 2 mg/day
  Interventions: Drug: Estradiol and Drospirenone

INTERVENTIONS:
Drug: Estradiol and Progesterone — 3 mg/day intranasal estradiol daily or 1,5 mg/day transdermal estradiol and 200 mg/day vaginal micronized progesterone for 14 days/month
  Arms: Non-oral hormone therapy
Drug: Estradiol and Drospirenone — oral estradiol 1mg and drospirenone 2 mg/day
  Arms: oral homone therapy

SUMMARY:
This is cross-over, randomized clinical trial, with objective to evaluate the effects of low-dose oral hormone therapy and non-oral hormone therapy on endothelial function markers (fibrinogen, von Willebrand factor, c-reactive protein), natriuretic peptide and on anthropometric, metabolic and hormonal variables in early and healthy postmenopausal women and analyzing polymorphisms in the estrogen receptor gene and FTO polymorphisms

Patients will be randomized to receive oral hormone treatment or non-oral hormone treatment

The investigators hypothesis is that a different genotypes in the receptor estrogen gene and FTO may have an influences on treatment response in metabolic markers and cardiovascular risk

ELIGIBILITY:
Inclusion criteria:

* last menstrual period between 6 months and 3 years before the beginning of the study plus FSH levels higher than 35 IU/L;
* age between 42 and 58 years;
* no use of any medication known to interfere with hormonal, glucose, or lipoprotein levels in the past 3 months;
* no use of steroidal or no steroidal anti-inflammatory drugs in the last 15 days.

Exclusion criteria:

* patients with diabetes,
* previous hysterectomy,
* endometrial thickness >0.5cm,
* history of cancer,
* thromboembolism, or
* established cardiovascular disease

Ages: 42 Years to 58 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2007-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Polymorphisms of estrogen receptor | six months
  Influence of 4 polymorphisms (PVUII, ALUI, RSAI and BSTUI) on the effect of different treatment regimens. Change from Baseline in weight, waist circumference, BMI, systolic and diastolic blood pressure, fasting glucose, glucose at 120 min, Fasting insulin, HOMA, Cholesterol, HDL-c, LDL-c, Triglycerides, Von Willebrand Factor, Fibrinogen, Testosterone and C-reactive protein at six months.

SECONDARY OUTCOMES:
Polymorphisms in the fat mass-and obesity-associated (FTO) gene | Six Months
  Influence of 2 polymorphisms (rs9939609 and rs8050136) on the effect of different treatment regimens. Change from Baseline in weight, waist circumference, BMI, systolic and diastolic blood pressure, fasting glucose, glucose at 120 min, Fasting insulin,HOMA, Cholesterol, HDL-c, LDL-c, Triglycerides, Von Willebrand Factor, Fibrinogen, Testosterone and C-reactive protein at six months.

OTHER OUTCOMES:
Effects of hormone therapy on C reactive protein, atrial natriuretic peptide and cardiovascular risk factors in postmenopause. | Six months
  To assess the effects of oral low-dose and non-oral hormone therapy (HT) on ultra-sensitive C reactive protein (CRP), atrial natriuretic peptide (ANP), and cardiovascular risk factors in postmenopause.

CONTACTS AND LOCATIONS:
Overall Officials: Poli Mara Spritzer, MD, PhD, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Casanova G, dos Reis AM, Spritzer PM. Low-dose oral or non-oral hormone therapy: effects on C-reactive protein and atrial natriuretic peptide in menopause. Climacteric. 2015 Feb;18(1):86-93. doi: 10.3109/13697137.2014.940309. Epub 2014 Oct 21. PMID 25017924
- [Derived] Casanova G, Spritzer PM. Effects of micronized progesterone added to non-oral estradiol on lipids and cardiovascular risk factors in early postmenopause: a clinical trial. Lipids Health Dis. 2012 Oct 9;11:133. doi: 10.1186/1476-511X-11-133. PMID 23046709
- [Derived] Ramos RB, Casanova GK, Spritzer PM. Fat mass and obesity-associated gene polymorphisms do not affect metabolic response to hormone therapy in healthy postmenopausal women. Eur J Obstet Gynecol Reprod Biol. 2012 Dec;165(2):302-6. doi: 10.1016/j.ejogrb.2012.07.024. Epub 2012 Aug 15. PMID 22901973